CLINICAL TRIAL: NCT03225833
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 1b/2a Study of WVE-120101 Administered Intrathecally in Patients With Huntington's Disease
Brief Title: Safety and Tolerability of WVE-120101 in Patients With Huntington's Disease
Acronym: PRECISION-HD1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-HDSNP1-001
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WVE-120101 (Dose A) or placebo (Experimental)
  Interventions: Drug: WVE-120101; Drug: Placebo
- WVE-120101 (Dose B) or placebo (Experimental)
  Interventions: Drug: WVE-120101; Drug: Placebo
- WVE-120101 (Dose C) or placebo (Experimental)
  Interventions: Drug: WVE-120101; Drug: Placebo
- WVE-120101 (Dose D) or placebo (Experimental)
  Interventions: Drug: WVE-120101; Drug: Placebo
- WVE-120101 (Dose E) or placebo (Experimental)
  Interventions: Drug: WVE-120101; Drug: Placebo

INTERVENTIONS:
Drug: WVE-120101 — WVE-120101 is a stereopure antisense oligonucleotide (ASO)
Drug: Placebo — 0.9% Sodium Chloride

SUMMARY:
PRECISION-HD1 is a Phase 1b/2a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple doses of WVE-120101 in adult patients with early manifest Huntington's disease (HD) who carry a targeted single nucleotide polymorphism (SNP) rs362307 (SNP1).

ELIGIBILITY:
Key Inclusion Criteria:

* Prescreened with targeted SNP on the same allele as the pathogenic CAG expansion
* Ambulatory, male or female patients aged ≥25 - ≤65 years
* Clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score = 4
* Early manifest HD, Stage I or Stage II based on UHDRS Total Functional Capacity Scores ≥7 and ≤13

Key Exclusion Criteria:

* Malignancy or received treatment for malignancy, other than treated basal cell or squamous cell carcinoma of the skin, within the previous 5 years.
* Received investigational drug or implantable device in prior 3 months or investigational oligonucleotide in prior 6 months or 5 half-lives of the oligonucleotide, whichever is longer
* Clinically significant medical condition, unstable psychiatric symptoms, substance abuse, or pregnancy
* Inability to undergo brain MRI
* Bone, spine, bleeding, or other disorder that exposes the patient to risk of injury or unsuccessful lumbar puncture

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (21):
- Australia (7):
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Melbourne Hospital, Carlton, Victoria
  - Monash Health, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria
  - Calvary Health Care Bethlehem, Parkdale, Victoria
  - North Metropolitan Health Service, Perth, Western Australia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Centre For Movement Disorders, Toronto, Ontario
  - Center Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Denmark (3):
  - Aarhus Universitets Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital and University of Southern Denmark, Odense
- France (2):
  - Hospital Henri Mondor, Créteil
  - Institut du Cerveau et de la Moelle Epinière, Paris
- George-Huntington-Institut GmbH, Münster, Germany
- Poland (2):
  - Szpital Sw. Wojciecha, Gdansk
  - Instytut Psychiatrii i Neurologii, Warsaw
- United Kingdom (3):
  - Royal Devon and Exeter Hospital NHS Trust, Exeter, Devon
  - Queen Elizabeth University Hospital - PPDS, Glasgow, Glasgow City
  - Royal Liverpool University Hospital, Liverpool

REFERENCES:
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: April 2020. J Huntingtons Dis. 2020;9(2):185-197. doi: 10.3233/JHD-200002. PMID 32250312
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: February 2018. J Huntingtons Dis. 2018;7(1):89-98. doi: 10.3233/JHD-189001. PMID 29480210

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: Placebo: 0.9% Sodium Chloride
- WVE-120101 (2 mg); WVE-120101 (4 mg); WVE-120101 (8 mg); WVE-120101 (16 mg); WVE-120101 (32 mg): WVE-120101: WVE-120101 is a stereopure antisense oligonucleotide (ASO)
Period: Overall Study
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Started | 16 | 9 | 9 | 9 | 8 | 10
Single Dose Period Only | 1 | 1 | 2 | 0 | 0 | 4
Multiple Dose Period Only | 0 | 0 | 0 | 0 | 0 | 1
Single Dose and Multiple Dose Periods | 15 | 8 | 7 | 9 | 8 | 5
Completed | 11 | 8 | 7 | 9 | 7 | 0
Not Completed | 5 | 1 | 2 | 0 | 1 | 10
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Termination of Study by Sponsor | 4 | 0 | 0 | 0 | 0 | 7
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg) | Total
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 9 | 9 | 9 | 8 | 10 | 60
  >=65 years | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 5 | 6 | 1 | 7 | 29
  Male | 9 | 6 | 4 | 3 | 7 | 3 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 9 | 9 | 9 | 8 | 10 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 16 | 9 | 9 | 9 | 8 | 10 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 2 | 2 | 1 | 0 | 3 | 12
  Denmark | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Poland | 4 | 7 | 5 | 1 | 2 | 0 | 19
  Australia | 4 | 0 | 0 | 6 | 3 | 4 | 17
  France | 1 | 0 | 0 | 0 | 1 | 2 | 4
  Germany | 2 | 0 | 0 | 0 | 1 | 1 | 4
  United Kingdom | 1 | 0 | 2 | 0 | 0 | 0 | 3
Time since initial diagnosis [Mean (Standard Deviation); unit: Years] | 7 (6.93) | 4.9 (4.28) | 3.4 (6.37) | 3.2 (3.03) | 6.6 (6.09) | 8.7 (7.26) | 5.4 (5.80)
Age at Disease Onset [Mean (Standard Deviation); unit: Years] | 40.75 (11.079) | 37.33 (7.826) | 42.89 (9.280) | 46.11 (6.254) | 44.88 (12.495) | 44.60 (10.865) | 43.16 (9.625)
Diagnosis Stage [Count of Participants; unit: Participants] — Stage of disease, as defined by United Huntington's Disease Rating Scale, Total Functional Capacity Score. Stage 1 (least severe) = scores of 11 to 13. Stage 2 = scores of 7 to 10. Stages go up to Stage 5 = score of 0.
  Participants
    Stage 1 | 9 | 7 | 3 | 3 | 4 | 7 | 33
    Stage 2 | 7 | 2 | 6 | 6 | 4 | 3 | 28

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Patients With Treatment-emergent Adverse Events (TEAEs)
Description: All TEAEs reported or observed during the study, including TEAEs resulting from concurrent illnesses, reactions to concurrent medications, or progression of disease states
Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10
Participants | 12 | 8 | 8 | 9 | 7 | 9

2. Primary Outcome: Safety: Severity of Adverse Events
Description: Number of patients who experienced a severe treatment-emergent adverse event. Severity was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10
Participants | 1 | 2 | 1 | 1 | 0 | 5

3. Primary Outcome: Safety: Number of Patients With Serious TEAEs
Description: A serious TEAE is defined as any event that results in death, is immediately life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect not present at Prescreening.
Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10
Participants | 0 | 2 | 1 | 0 | 0 | 4

4. Primary Outcome: Safety and Tolerability: Number of Patients Who Withdraw Due to TEAEs
Time Frame: Day 1 to end of study (up to Day 182 [32 mg cohort]/ Day 210 [all other cohorts])
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10
Participants | 0 | 1 | 2 | 0 | 0 | 2

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax)
Description: Cmax of WVE-120101 in plasma
Time Frame: Patients participating in Period 1 (SAD) had PK samples collected on Day 1 predose through 24-48 hours postdose. Patients participating in Period 2 (MAD) had PK samples collected predose on Day 112 and through 4 hours postdose.
Population: The PK population consists of all treated patients in the safety population with at least 1 post-dose plasma or CSF WVE-120101 concentration measurement. The number of overall participants analyzed represents the number with at least 1 postdose plasma or CSF measurement at Day 1. The overall number of patients was different for Day 112, and represents patients with at least 1 postdose plasma or CSF measurement at Day 112.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
ng/mL
  Day 1 | 7.70 (7.901) | 23.54 (18.139) | 32.82 (22.964) | 184.48 (209.470) | 229.01 (168.330)
  Day 112: number analyzed (Participants) | 8 | 4 | 0 | 0 | 0
  Day 112 | 13.296 (6.057) | 14.27 (12.574) |  |  |

6. Secondary Outcome: PK: Time of Occurrence of Cmax (Tmax)
Description: tmax of WVE-120101 in plasma
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
hours
  Day 1 | 1.34 (1.103) | 1.58 (1.081) | 2.66 (1.391) | 2.71 (3.068) | 4.61 (7.054)
  Day 112: number analyzed (Participants) | 8 | 4 | 0 | 0 | 0
  Day 112 | 1.99 (0.934) | 2.23 (1.175) |  |  |

7. Secondary Outcome: PK: Area Under the Plasma Concentration-time Curve (AUClast)
Description: AUClast from time 0 to the last quantifiable concentration of WVE-120101 in plasma
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
hr*ng/mL
  Day 1 | 35.20 (16.037) | 90.77 (50.672) | 255.14 (98.342) | 1133.74 (551.997) | 1968.31 (1188.173)
  Day 112: number analyzed (Participants) | 8 | 4 | 0 | 0 | 0
  Day 112 | 36.19 (20.135) | 49.54 (34.735) |  |  |

8. Secondary Outcome: PK: Terminal Elimination Half Life
Description: Terminal elimination half life of WVE-120101 in plasma (t1/2)
Time Frame: as for outcome 5
Population: The t1/2 value was calculated using data from patients who had at least 3 postdose concentration values in the terminal phase. No patients had sufficient postdose samples at Day 112 to calculate t1/2 values.
Measure: Median (Full Range); unit: hours
Arm/Group | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 0 | 0 | 3 | 3 | 6
hours |  |  | 8.12 [7.1 to 40.0] | 12.30 [6.9 to 25.5] | 14.38 [5.5 to 46.9]

9. Secondary Outcome: Pharmacodynamics
Description: Percentage change from baseline in concentration of mutant huntingtin (mHTT) protein in CSF
Time Frame: Day 1 to last observation - up to Day 140 (32 mg cohort) or Day 196 (all other cohorts)
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10
Percent change from baseline | -6.62 [-16.76 to 7.73] | -5.20 [-10.94 to 0.15] | -12.33 [-19.81 to 9.63] | -8.58 [-11.92 to -1.79] | -11.73 [-20.44 to 3.37] | -9.13 [-37.51 to 15.29]

10. Secondary Outcome: Clinical Effects: Total Functional Capacity (TFC)
Description: Percentage change from baseline to the last measured time point in the Total Functional Capacity score, administered as part of the Unified Huntington's Disease Rating Scale (UHDRS). Total Functional Capacity is scored 13 (normal) to 0 (severe disability).
Time Frame: Day 1 to last observation - up to Day 140 (32 mg cohort) or Day 196 (all other cohorts)
Measure: Median (Inter-Quartile Range); unit: % Change from Baseline
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
Number analyzed (Participants) | 16 | 9 | 9 | 9 | 8 | 10
% Change from Baseline | 0.00 [-9.09 to 0.00] | 0.00 [-4.17 to 9.09] | 0.00 [-7.69 to 11.11] | 0.00 [-20.00 to 0.00] | 4.17 [-3.85 to 10.42] | 0.00 [0.00 to 0.00]

ADVERSE EVENTS:
Time Frame: Day 1 to end of study (Day 196 [32 mg cohort] or Day 210 [all other cohorts])
Arm/Group | Pooled Placebo | WVE-120101 (2 mg) | WVE-120101 (4 mg) | WVE-120101 (8 mg) | WVE-120101 (16 mg) | WVE-120101 (32 mg)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/9 | 0/9 | 0/9 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/9 | 1/9 | 0/9 | 0/8 | 4/10
Other Adverse Events (participants affected / at risk) | 12/16 | 8/9 | 8/9 | 9/9 | 7/8 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=16) | WVE-120101 (2 mg) (N=9) | WVE-120101 (4 mg) (N=9) | WVE-120101 (8 mg) (N=9) | WVE-120101 (16 mg) (N=8) | WVE-120101 (32 mg) (N=10)
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=16) | WVE-120101 (2 mg) (N=9) | WVE-120101 (4 mg) (N=9) | WVE-120101 (8 mg) (N=9) | WVE-120101 (16 mg) (N=8) | WVE-120101 (32 mg) (N=10)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Administration site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Administration site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 3 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 2 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
CSF lymphocyte count increase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
CSF protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
CSF white blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 2 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 1 | 2 | 2 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Chorea (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Hyperreflexia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pleocytosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Radicular pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 1 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03225833/Prot_SAP_000.pdf